CLINICAL TRIAL: NCT06263972
Title: Comparison of the Efficacy of Transcranial Direct Current Stimulation (tDCS) of the Primary Motor Cortex (M1) or the Prefrontal Cortex Combined With Aerobic Activity for Alleviation of Fibromyalgia Symptoms and on Improving Self-Regulation and Quality of Life- a Randomized, Double Blinded Controlled Prospective Study
Brief Title: Comparison of the Efficacy of Transcranial Direct Current Stimulation (tDCS) of the Primary Motor Cortex (M1) or the Prefrontal Cortex Combined With Aerobic Activity for Alleviation of Fibromyalgia Symptoms.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shahak Yariv, Doctor, Head of neuromodulation, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0168-21EMC
Record Dates: First submitted 2023-12-11; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia; Electric Shock
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Stimulation of the Primary Motor Cortex (M1) Combined With Aerobic Activity. (Active Comparator): low current electrical stimulation to Motor cortex for 3 weeks.
  Interventions: Device: Direct Stimulation to Motor Cortex; Behavioral: erobic physical activity
- Direct Stimulation the Prefrontal Cortex Combined With Aerobic Activity (Active Comparator): with low current electrical stimulation to Prefrontal cortex for 3 weeks.
  Interventions: Device: Direct Stimulation Prefrontal Cortex; Behavioral: erobic physical activity
- Shame Stimulation Combined With Aerobic Activity (Sham Comparator): Shame low current electrical stimulation to cortex for 3 weeks.
  Interventions: Device: Shame cortex stimulation; Behavioral: erobic physical activity

INTERVENTIONS:
Device: Direct Stimulation Prefrontal Cortex — The therapeutic course will include moderate aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment), along with low current electrical stimulation to prefrontal cortex for 3 weeks.
  Arms: Direct Stimulation the Prefrontal Cortex Combined With Aerobic Activity
Device: Shame cortex stimulation — The therapeutic course will include moderate aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment), along with shame low current electrical stimulation to cortex for 3 weeks.
  Arms: Shame Stimulation Combined With Aerobic Activity
Device: Direct Stimulation to Motor Cortex — The therapeutic course will include moderate aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment), along with low current electrical stimulation to Motor cortex for 3 weeks.
  Arms: Direct Stimulation of the Primary Motor Cortex (M1) Combined With Aerobic Activity.
Behavioral: erobic physical activity — Aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment),

SUMMARY:
The goal of this study is to demonstrate the effectiveness of treating fibromyalgia using combination of electrical stimulation with aerobic activity.

Participants will be randomly assigned to stimulation in a ratio of 1:1:1. 120 participants (40 in each group). The therapeutic course will include moderate aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment), along with low current electrical stimulation for 3 weeks.

DETAILED DESCRIPTION:
Fibromyalgia is a disorder of unknown origin that causes widespread pain, fatigue, sleep disorders, cognitive disorders, depression and anxiety. Today, the treatments for fibromyalgia are limited in their effectiveness in most cases. Previous works have demonstrated that the self-regulation ability among those dealing with fibromyalgia is impaired, and their quality of life is poor.

Therapy using low current electrical stimulation is considered an effective, safe and non-invasive means of treating various disorders including treatment of depression, neurological rehabilitation and various pain syndromes.

A number of works have demonstrated the effectiveness of treating fibromyalgia using stimulation using low electrical current , and it has also been demonstrated that a combination of electrical stimulation with aerobic activity improved the results, together with each of the treatments separately. There are several areas that can be stimulated including the primary motor area (M1) and the prefrontal area , however, the studies performed were limited to a relatively small number of subjects, and no direct comparison was made between the different stimulation locations.

For the study, male and female patients dealing with fibromyalgia will be recruited from the hospital clinics or those who will be referred by the attending physician, or will respond to recruitment notices, in total we intend to recruit 120 participants (40 in each group). The patients will be randomly assigned to real stimulation for each of the areas or to blood stimulation in a ratio of 1:1:1. The therapeutic course will include moderate aerobic physical activity (at 60% of the target heart rate adjusted for age) 3 times a week for 4 weeks (a week of adjustment, and 3 weeks of treatment), along with low current electrical stimulation for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Fibromyalgia
* Pain scale level of 4 or higher
* Fail to achieve adequate pain relief with Fibromyalgia treatments
* stable Fibromyalgia treatment for at least 4 weeks.
* Ability to perform aerobic exercise

Exclusion Criteria:

* Other Causes of pain
* Psychotic disorder
* Severe Depression
* Cognitive disorder
* Drug or alcohol abuse in the last 6 months
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Study objectives: • Comparing the effectiveness of direct electric current stimulation between the two stimulus areas Numeric pain rating scale. | 3 months
  Study objectives:
  • Comparing the effectiveness of direct electric current stimulation (tDCS) between the two stimulus areas and in relation to blood stimulation.
  Based on:
  Numeric pain rating scale (score range from 1 to 10)
Study objectives: • Comparing the effectiveness of direct electric current stimulation (tDCS) between the two stimulus areas and in relation Adult sensory profile test Raw score. | 3 months
  Study objectives:
  • Comparing the effectiveness of direct electric current stimulation (tDCS) between the two stimulus areas and in relation to blood stimulation.
  Based on:
  Adult sensory profile test Raw score
Study objectives: • Comparing the effectiveness of direct electric current stimulation between the two stimulus areas and in relation to The Montreal Cognitive Assessment (MoCA) score. | 3 months
  Study objectives:
  • Comparing the effectiveness of direct electric current stimulation (tDCS) between the two stimulus areas and in relation to The Montreal Cognitive Assessment (MoCA) score.
  Based on:
  The Montreal Cognitive Assessment (MoCA) score
Study objectives: • Comparing the effectiveness of direct electric current stimulation between the two stimulus areas and in relation to Generalized Anxiety Disorder 7-Item Scale | 3 months
  Study objectives:
  • Comparing the effectiveness of direct electric current stimulation (tDCS) between the two stimulus areas and in relation to blood stimulation.
  Based on:
  The Generalized Anxiety Disorder 7-Item Scale

IPD SHARING:
Plan to Share IPD: No